CLINICAL TRIAL: NCT03366480
Title: A Phase I/II, Open Label Study to Assess the Efficacy and Safety of ABTL0812 in Combination With Paclitaxel and Carboplatin in Patients With Advanced Endometrial Cancer or Squamous NSCLC
Brief Title: A Study to Assess the Efficacy and Safety of ABTL0812
Acronym: Endolung
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ability Pharmaceuticals SL (Industry)
Collaborators: Hospital Vall d'Hebron (Other); Institut Català d'Oncologia (Other); Hospital Clínico Universitario de Valencia (Other); Hospitales Universitarios Virgen del Rocío (Other); Centre Leon Berard (Other); Institut Paoli-Calmettes (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-C5-2016; 2016-001352-21 (EudraCT Number)
Record Dates: First submitted 2017-11-15; First posted 2017-12-08 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Endometrial Cancer; Squamous Non-Small Cell Lung Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ABTL0812; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial cancer (Experimental): ABTL0812 (starting 1,300 mg tid orally) in combination with paclitaxel and carboplatin will be given to patients with advanced endometrial cancer, up to 12 months from initiation.
  Interventions: Drug: ABTL0812 in combination with paclitaxel and carboplatin
- Squamous non-small cell lung cancer (Experimental): ABTL0812 (starting 1,300 mg tid orally) in combination with paclitaxel and carboplatin will be given to patients with squamous NSCLC, up to 12 months from initiation.
  Interventions: Drug: ABTL0812 in combination with paclitaxel and carboplatin

INTERVENTIONS:
Drug: ABTL0812 in combination with paclitaxel and carboplatin — ABTL0812 in combination with paclitaxel and carboplatin.

SUMMARY:
A phase I/ II, open label study to assess the efficacy and safety of ABTL0812 in combination with paclitaxel and carboplatin in patients with advanced endometrial cancer or squamous NSCLC.

DETAILED DESCRIPTION:
This is a phase I/II multicenter divided in two phases.

Phase I: Safety and dose escalation

This study is not randomized, and all included patients will receive ABTL0812 in addition to paclitaxel + carboplatin (SOC). In this phase, patients can be selected from both indications, regardless of the number of each indication.

This phase will be divided in 2 periods:

Period 1:

A dose de-escalation phase will be performed with a 3 + 3 design, in which up to four different ABTL0812 dose levels will be tested in combination with SOC. Then, 12 patients will be included in an expansion phase. All patients will receive one week of ABTL0812 alone followed by ABTL0812 + SOC (up to 8 SOC cycles) as combined treatment.

Period 2:

After the finalization of the SOC cycles, ABTL0812 will be taken as single therapy, at 1300 mg tid, up to 12 months from initiation of period 1. This is the Recommended Phase 2 Dose (RP2D) as monotherapy for ABTL0812 determined in the previous phase I clinical trial.

Phase II: Efficacy and safety

This phase of the study will include up to 33 patients per indication (up to 66 patients overall). The final number will depend on the number of patients included in the phase I. The number of patients selected per indication will depend on the number already selected in phase I, as it is necessary to compensate both indications to have a final number of 40 patients per indication approximately.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Willing and able to provide informed consent
* For endometrial cancer: Patients with advanced, metastatic or recurrent endometrial cancer, from all histological types except carcinosarcoma and leiomyosarcoma.
* For squamous NSCLC: Patients with histologically or radiological/cytologically confirmed diagnosis (non-irradiance IIIb stage or stage IV), excluding mixed tumors, neuroendocrine or adenocarcinoma.
* Have adequate tumor tissue available (either archival not older than 6 months or new tumor biopsy) for biomarker analyses. The most recently collected tumor tissue sample should be provided, if available.
* Life expectancy ≥ 12 weeks in the opinion of the investigator
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 guidelines with at least one "target lesion" to be used to assess response. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Contraception: All female patients will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months' consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically. Female patients of childbearing potential must agree to use two forms of highly effective contraception methods during the study and for a period of 6 months following the last administration of the study drug. Male patients and their female partners, who are of childbearing potential and are not practicing total abstinence, must agree to use two forms of highly effective contraception during the study and for a period of 6 months following the last administration of the study drug.
* Adequate bone marrow function defined as:

  * absolute neutrophil count ≥ 1.5x109/L
  * platelet count ≥ 100x109/L
  * hemoglobin ≥ 10.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal
* Aspartate transaminase (AST) ≤ 2.5 times upper limit of normal (ULN) (≤5 times the ULN in patients with evidence of liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN (≤5 times the ULN in patients with evidence of liver metastases)
* Glomerular filtration rate ≥ 50 mL/min
* Serum creatinine ≤1.5 ULN
* Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 1 (as defined by Common Terminology Criteria for Adverse Events version 4.02).
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol

Exclusion Criteria:

* Patients previously treated with an inhibitor of the Phosphoinositide 3-kinase/Protein kinase B/mechanistic target of rapamycin (PI3K/Akt/mTOR) pathway.
* Patients previously treated with adjuvant or co-adjuvant chemotherapy administered 6 months or less in advance of patient inclusion
* Patients with symptomatic brain metastases. Patients with asymptomatic and treated brain metastases can be included in the study if they are kept on stable doses of steroids for a period of 1 month prior to study entry provided they don't have peripheric neuropathy grade 2 or superior.
* Patients with gastrointestinal abnormalities including inability to take oral medications, malabsorption syndromes or other clinically significant gastrointestinal abnormalities that may impair the absorption of the investigational medicinal product.
* Pregnancy or lactation. Serum pregnancy test to be performed within 7 days prior to study treatment start.
* Patients with myocardial infarction within ≤ 12 months prior to study entry, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina pectoris, or unstable cardiac arrhythmia requiring medication.
* Evidence of pre-existing uncontrolled hypertension. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Patients with active Hepatitis B or C or human immunodeficiency virus (HIV) infection with non-controlled disease according to the treating physician.
* Patients with any other medical conditions (such as psychiatric illness, infectious diseases, abnormal physical examination or laboratory findings) that in the opinion of the investigator may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Emergent Adverse Events | 1 year
  Related Adverse Events as Assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Objective response rate (ORR) based on tumor assessment by CT-Scan according to RECIST criteria version 1.1. performed at baseline and at every other treatment visit, starting at 3rd SOC cycle
Progression Free Survival (PFS) | 2 years
  Progression Free Survival (PFS) based on tumor assessment by CT-Scan according to RECIST criteria version 1.1. performed at baseline and at every other treatment visit, starting at 3rd SOC cycle
Time to Progression (TP) | 2 years
  Time to Progression (TP) based on tumor assessment by CT-Scan according to RECIST criteria version 1.1. performed at baseline and at every other treatment visit, starting at 3rd SOC cycle
Duration of Response (DR) | 2 years
  Duration of Response (DR), based on tumor assessment by CT-Scan according to RECIST criteria version 1.1. performed at baseline and at every other treatment visit, starting at 3rd SOC cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, Principal Investigator — VHIO
Locations (1):
- Abilitypharma, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erazo T, Lorente M, Lopez-Plana A, Munoz-Guardiola P, Fernandez-Nogueira P, Garcia-Martinez JA, Bragado P, Fuster G, Salazar M, Espadaler J, Hernandez-Losa J, Bayascas JR, Cortal M, Vidal L, Gascon P, Gomez-Ferreria M, Alfon J, Velasco G, Domenech C, Lizcano JM. The New Antitumor Drug ABTL0812 Inhibits the Akt/mTORC1 Axis by Upregulating Tribbles-3 Pseudokinase. Clin Cancer Res. 2016 May 15;22(10):2508-19. doi: 10.1158/1078-0432.CCR-15-1808. Epub 2015 Dec 15. PMID 26671995
- [Background] Munoz-Guardiola P, Casas J, Megias-Roda E, Sole S, Perez-Montoyo H, Yeste-Velasco M, Erazo T, Dieguez-Martinez N, Espinosa-Gil S, Munoz-Pinedo C, Yoldi G, Abad JL, Segura MF, Moran T, Romeo M, Bosch-Barrera J, Oaknin A, Alfon J, Domenech C, Fabrias G, Velasco G, Lizcano JM. The anti-cancer drug ABTL0812 induces ER stress-mediated cytotoxic autophagy by increasing dihydroceramide levels in cancer cells. Autophagy. 2021 Jun;17(6):1349-1366. doi: 10.1080/15548627.2020.1761651. Epub 2020 May 25. PMID 32397857
- [Background] Felip I, Moiola CP, Megino-Luque C, Lopez-Gil C, Cabrera S, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Alfon J, Yeste-Velasco M, Santacana M, Dolcet X, Reques A, Oaknin A, Rodriguez-Freixinos V, Lizcano JM, Domenech C, Gil-Moreno A, Matias-Guiu X, Colas E, Eritja N. Therapeutic potential of the new TRIB3-mediated cell autophagy anticancer drug ABTL0812 in endometrial cancer. Gynecol Oncol. 2019 May;153(2):425-435. doi: 10.1016/j.ygyno.2019.03.002. Epub 2019 Mar 7. PMID 30853360
- [Background] Lopez-Plana A, Fernandez-Nogueira P, Munoz-Guardiola P, Sole-Sanchez S, Megias-Roda E, Perez-Montoyo H, Jauregui P, Yeste-Velasco M, Gomez-Ferreria M, Erazo T, Ametller E, Recalde-Percaz L, Moragas-Garcia N, Noguera-Castells A, Mancino M, Moran T, Nadal E, Alfon J, Domenech C, Gascon P, Lizcano JM, Fuster G, Bragado P. The novel proautophagy anticancer drug ABTL0812 potentiates chemotherapy in adenocarcinoma and squamous nonsmall cell lung cancer. Int J Cancer. 2020 Aug 15;147(4):1163-1179. doi: 10.1002/ijc.32865. Epub 2020 Feb 6. PMID 31943158
- [Background] Vidal L, Victoria I, Gaba L, Martin MG, Brunet M, Colom H, Cortal M, Gomez-Ferreria M, Yeste-Velasco M, Perez A, Rodon J, Sohal DPS, Lizcano JM, Domenech C, Alfon J, Gascon P. A first-in-human phase I/Ib dose-escalation clinical trial of the autophagy inducer ABTL0812 in patients with advanced solid tumours. Eur J Cancer. 2021 Mar;146:87-94. doi: 10.1016/j.ejca.2020.12.019. Epub 2021 Feb 12. PMID 33588149
- [Background] Paris-Coderch L, Soriano A, Jimenez C, Erazo T, Munoz-Guardiola P, Masanas M, Antonelli R, Boloix A, Alfon J, Perez-Montoyo H, Yeste-Velasco M, Domenech C, Roma J, Sanchez de Toledo J, Moreno L, Lizcano JM, Gallego S, Segura MF. The antitumour drug ABTL0812 impairs neuroblastoma growth through endoplasmic reticulum stress-mediated autophagy and apoptosis. Cell Death Dis. 2020 Sep 17;11(9):773. doi: 10.1038/s41419-020-02986-w. PMID 32943619
- [Background] Mancini A, Colapietro A, Cristiano L, Rossetti A, Mattei V, Gravina GL, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Domenech C, Festuccia C. Anticancer effects of ABTL0812, a clinical stage drug inducer of autophagy-mediated cancer cell death, in glioblastoma models. Front Oncol. 2022 Nov 2;12:943064. doi: 10.3389/fonc.2022.943064. eCollection 2022. PMID 36408162
- [Derived] Leary A, Estevez-Garcia P, Sabatier R, Ray-Coquard I, Romeo M, Barretina-Ginesta P, Gil-Martin M, Garralda E, Bosch-Barrera J, Moran T, Martin-Martorell P, Nadal E, Gascon P, Rodon J, Lizcano JM, Munoz-Guardiola P, Fierro-Duran G, Pedros-Gamez O, Perez-Montoyo H, Yeste-Velasco M, Cortal M, Perez-Campos A, Alfon J, Domenech C, Perez-Fidalgo A, Oaknin A. ENDOLUNG trial. A phase 1/2 study of the Akt/mTOR inhibitor and autophagy inducer Ibrilatazar (ABTL0812) in combination with paclitaxel/carboplatin in patients with advanced/recurrent endometrial cancer. BMC Cancer. 2024 Jul 22;24(1):876. doi: 10.1186/s12885-024-12501-5. PMID 39039449
- [Derived] Polonio-Alcala E, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Lizcano JM, Domenech C, Ruiz-Martinez S, Puig T. ABTL0812 enhances antitumor effect of paclitaxel and reverts chemoresistance in triple-negative breast cancer models. Cancer Commun (Lond). 2022 Jun;42(6):567-571. doi: 10.1002/cac2.12282. Epub 2022 Mar 16. No abstract available. PMID 35293148